CLINICAL TRIAL: NCT03075202
Title: Role of an E-cigarette on Smoking Displacement in Smokers With Schizophrenia: A Prospective 3-month Pilot Study
Brief Title: Role of an E-cigarette on Smoking Displacement in Smokers With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hunter College of The City University of New York (Other); University of Catania (Other); University of Stirling (Other)
Responsible Party: Sponsor
Other Study IDs: 1607017418
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia; Smoking; E-cigarette
MeSH Terms: conditions — Schizophrenia; Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: e-cigarette, brand name JUUL — This is not an experimental study/trial, rather a prospective observational study. Device will be offered to cohort, but they are not mandated to take or use the device.

SUMMARY:
It is well established in the scientific literature that people with schizophrenia smoke tobacco cigarettes at rates up to three times that of the general population, relapse more frequently, and die an average of 25 years earlier from cigarette smoking and other life-style attributable illnesses. Electronic cigarettes (e-cigarettes) are becoming increasingly popular with smokers worldwide and new research suggests that e-cigarettes are appealing to smokers with schizophrenia. There is a paucity of research focused on the experience of smokers with schizophrenia who decide to try an e-cigarette. A well-designed prospective-observational study is needed to learn more about the influence of e-cigarette use on cigarette smoking behavior and mental and physical health among smokers with schizophrenia. In response, the investigators have designed a study titled, Role of an electronic cigarette on smoking displacement in smokers with schizophrenia: A prospective 3-month pilot study (SchizEcig).

DETAILED DESCRIPTION:
This is a prospective 3 month pilot study to observe cigarette use behavior among people with a schizophrenia spectrum disorder diagnosis who smoke conventional tobacco cigarettes, do not intend to reduce or quit smoking, and are invited to use an e-cigarette. The investigators are interested to know if e-cigarette use is associated with cigarette smoking displacement. Displacement is defined as switching from conventional tobacco cigarettes to e-cigarettes. The investigators will also monitor for physical and mental health, including blood pressure, weight, and scores from the Scale for the Assessment of Negative Symptoms (SANS) and the Scale for the Assessment of Positive Symptoms (SAPS) as well as any reported adverse events participants' feel are attributed to e-cigarette use and participants' perceptions of the sensory experience associated with e-cigarette use.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of a schizophrenia spectrum disorder

Non-hospitalized persons

Regular smokers who report smoking 20 or more cigarettes per day who have smoked at least 100 cigarettes in their lifetime, and are not intending to reduce or quit

Has agreed to try an e-cigarette

Must be able to provide written informed consent

Must be able to read, write and communicate in English proficiently

Must have access to a computer with internet

Must have the ability to work a computer and navigate the internet easily

Exclusion Criteria:

Non-smokers Persons without a schizophrenia spectrum disorder diagnosis

Hospitalized persons

Cardio vascular disease

Respiratory disease

Use of smokeless tobacco or any other tobacco products besides cigarettes.

Use of nicotine replacement therapy or other smoking cessation pharmaco-therapies within the last 3 months

Pregnancy or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants, age 21 to 65 years, will have a DSM 5 schizophrenia spectrum disorder diagnosis without evidence of exacerbation of illness as indicated by no relapse to hospitalization within the last three months and no change in their antipsychotic treatment within the last month. Participants will smoke 20 or more conventional tobacco cigarettes per day and at least 100 cigarettes in their lifetime and do not intend to reduce or quit smoking.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Smoking Displacement | 3-months
  The primary endpoint of this study is the proportion of study participants with a self-reported complete displacement from tobacco cigarette smoking - not even a puff in between study visits, along with confirmatory eCO values ≤10 ppm at each study visit. These participants will be referred to as "Displacers". Discrepancies between self-report and eCO measures will be handled on a case-by-case basis. To assure an accurate eCO reading participants will be asked not to smoke cigarettes within one hour of the study visit.

SECONDARY OUTCOMES:
Partial Displacement | 3-months
  Partial displacement will be defined as a minimization in cigarette consumption by ≥50% in the number of tobacco cigarettes smoked per day from baseline to the final visit (week 12) by participants' self-report together with an eCO decline from baseline.. The measures will be taken at each study visit. These participants will be referred to as "Partial Displacers". Discrepancies between self-report and eCO measures will be handled on a case-by-case basis. To assure an accurate eCO reading participants will be asked not to smoke cigarettes within one hour of the study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DiPiazza-Sileo, PhD, PMHNP, Principal Investigator — Hunter College at The City University of New York; Caponnetto Pasquale, PhD, Principal Investigator — University of Catania; Jason J Kim, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Clinical and Translational Science Center, Weill Cornell Medicine, 525 E 68th Street, F-260, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be available to some collaborating researchers, but not all.